CLINICAL TRIAL: NCT01416337
Title: Determination of the Absolute Bioavailability of GSK1120212 Following a Single Oral Dose Co-Administered With an Intravenous Radiolabelled Microdose of GSK1120212 in Subjects With Solid Tumors
Brief Title: Absolute Bioavialability of GSK1120212
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115064
Record Dates: First submitted 2011-08-11; First posted 2011-08-15 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatments A & B (Experimental): Single 2 mg GSK1120212 oral tablet, fasted Single IV dose of 5 ug (no more than 7.4 kBq or 200 nCi) [14C]GSK1120212 Both doses are given together.
  Interventions: Drug: GSK1120212; Drug: GSK1120212B

INTERVENTIONS:
Drug: GSK1120212 — 2 mg single dose tablet on Day 1 of study
Drug: GSK1120212B — A single administration of a slow 1 minute IV push on Day 1.

SUMMARY:
A Phase I, single-center, open-label, single-persiod, combined single dose oral and IV microtracer study in subjects with solid tumors.

DETAILED DESCRIPTION:
This Phase I, open-label, non-randomized study is designed to determine the absolute bioavailability of the standard 2 mg tablet formulation of GSK1120212 co-administered with an intravenous microdose (5 μg) dose of [14C]-labelled GSK1120212 (7.4 kBq) in subjects with solid tumors. Pharmacokinetic sampleswill be obtained up to 10 days post-dose. Safety assessments, including assessment of adverse events, clinical laboratory values (hematology and clinical chemistry) and vital signs, will be performed throughout the study. After completing all assessments, eligible subjects may transition to MEK114375, an open-label, rollover study to continue treatment with GSK1120212.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 18 years of age at the time of signing the informed consent form
2. Histologically or cytologically confirmed diagnosis of a solid tumor that is not responsive to standard therapies or for which there is no approved therapy.
3. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
4. Body weight greater than or equal to 45 kg and a body mass index greater than or equal to 19 kg/m2 and less than 35 kg/m2 (inclusive)
5. Able to swallow and retain oral medication
6. Has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
7. Women of child-bearing potential and men with reproductive potential must be willing to practice acceptable methods of birth control (see Section 7.1). Additionally, women of childbearing potential must have a negative serum pregnancy test within 14 days prior to the first dose of study treatment;
8. Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception as described in Section 7.1 from the time of first dose of study treatment until 16 weeks following the last dose of study treatment (based on the lifecycle of sperm).
9. Must have adequate organ function as defined in Table 4:

Table 4 Definitions for Adequate Baseline Organ Function System Laboratory Values Hematologic Absolute neutrophil count greater than or equal to 1.2 × 109/L Hemoglobin greater than or equal to 9 g/dL Platelets greater than or equal to 75 × 109/L Prothrombin time (PT), International normalization ratio (INR)a and Partial thromboplastin time (PTT) less than or equal to 1.5 times ULN Total bilirubin less than or equal to 1.5 times ULN ALT less than or equal to 2.5 times ULN Creatinine or less than or equal to 1.5 times ULN Calculated creatinine clearance b or greater than or equal to 50 mL/min 24-hour urine creatinine clearance greater than or equal to 50 mL/min LVEF greater than or equal to LLNc by ECHO or MUGA

1. INR greater1.5 times ULN will be acceptable in case of subjects receiving therapeutic anticoagulants such as warfarin as long as INR is monitored during the study according to clinical practice.
2. Calculated by the Cockcroft-Gault formula (see Appendix 4).
3. If LLN is not defined for a given institution, then ejection fraction must be greater than or equal to 50%. NOTE: Subjects with ALT or bilirubin values outside the range(s) in the table due to Gilbert's syndrome or asymptomatic gallstones are not excluded. Laboratory results obtained during Screening should be used to determine eligibility criteria. In situations where laboratory results are outside the permitted range, the investigator may opt to retest the subject and the subsequent within-range screening result may be used to confirm eligibility.

Exclusion Criteria:

1. Currently receiving cancer therapy (e.g., chemotherapy with delayed toxicity, extensive radiation therapy, immunotherapy, biologic therapy, or major surgery) within the last 3 weeks; chemotherapy regimens without delayed toxicity within the last 2 weeks; or use of an investigational anti-cancer drug within 28 days preceding dosing of GSK1120212; use of any other investigational product within 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (IP) (whichever is longest);
2. Has participated in a 14C human research study in the 12 months prior to administration of study treatment;
3. Current use of a prohibited medication (Section 8.2) or requires any of these medications during the study NOTE: Use of anticoagulants such as warfarin is permitted; however, INR must be monitored in accordance with local institutional practice.
4. Has unresolved Grade 2 or greater toxicity (based on NCI-CTCAE, version 4.0) [NCI, 2009] from previous anti-cancer therapy except alopecia and Grade 2 anemia level.
5. Has pre-existing Grade 2 or greater peripheral neuropathy.
6. Has participated in a study that resulted in or made a donation of blood or blood products in excess of 500 mL within 56 days of the first dose of study treatment.
7. Has presence of active GI disease or other condition (e.g., gastrectomy, bariatric surgery, small or large bowel resection, or cholecystectomy should be excluded) that may interfere significantly with the absorption of drugs. If clarification is needed as to whether a condition will significantly affect absorption of drugs, contact the GSK Medical Monitor.
8. Has any serious and/or unstable pre-existing medical (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures, in the opinion of the investigator or GSK Medical Monitor.
9. Has a history of interstitial lung disease or pneumonitis.
10. Has a history or current evidence/risk of RVO or CSR:

    * History of RVO or CSR, or predisposing factors to RVO or CSR (i.e., uncontrolled glaucoma or ocular hypertension, uncontrolled systemic disease such as hypertension or diabetes mellitus, or history of hyperviscosity or hypercoagulability syndromes)
    * Visible retinal pathology as assessed by ophthalmic exam that is considered a risk factor for

    RVO or CSR such as:
    * Evidence of new optic disc cupping
    * Intraocular pressure >21 mmHg as measured by tonography
11. Has symptomatic or untreated leptomeningeal or brain metastases or spinal cord compression.

    Note: Subjects previously treated for these conditions that have had stable central nervous system disease (verified with consecutive imaging studies) for >3 months, are asymptomatic and are not currently taking corticosteroids, or are on stable dose of corticosteroids for at least 1 month prior to Day 1 of the study are permitted.
12. QTcF (preferred) or QTcB greater than or equal to 480 msec.
13. Has a history or evidence of cardiovascular risk including any of the following:

    * History or evidence of current clinically significant uncontrolled arrhythmias. Exception:

Subjects with controlled atrial fibrillation for >30 days prior to enrollment are eligible.

* History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to enrollment.
* History or evidence of current ≥ Class II congestive heart failure as defined by New York Heart Association [NYHA, 1994] (Appendix 3) NOTE: Subjects with BBB are not excluded from this study; however, if the underlying cause of the BBB is exclusionary or if the BBB is new onset (therefore, potentially reflective of an evolving cardiac condition), the subject should be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-06-20 (Actual); Primary Completion 2011-12-17 (Actual); Study Completion 2011-12-17 (Actual)

PRIMARY OUTCOMES:
Determine the the absolute bioavailability of GSK1120212 following single oral tablet dose co-administered with an IV microdose. | Pre-dose, 0.5h, 1h, 1.5h, 1.55h, 1.75h,2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 10h, 24h, 48h, 72h, 120h, 168h, and 240h.
  Absolute bioavailability (F) of GSK1120212 calculated as the ratio of dose-normalized area under the concentration-time curve from time 0 (pre-dose) extrapolated to infinity (AUC(0-inf)) of oral to IV dosing

SECONDARY OUTCOMES:
Determine the single dose PK of GSK1120212 following oral administration. | Pre-dose, 0.5h, 1h, 1.5h, 1.75h,2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 10h, 24h, 48h, 72h, 120h, 168h, and 240h.
  Oral dosing: Cmax, tmax, AUC(0 24), area under the concentration-time curve from time 0 (pre-dose) to time t (AUC(0-t)), AUC(0-inf), t1/2, oral clearance (CL/F) of GSK1120212
Determine the single dose PK of GSK1120212 following IV administration. | 1.55h, 1.75h,2h, 2.5h, 3h, 4h, 5h, 6h, 8h, 10h, 24h, 48h, 72h, 120h, 168h, and 240h.
  IV dosing: Cmax, tmax, AUC(0-24), AUC(0-t), AUC(0-inf), t1/2, systemic clearance (CL), and volume of distribution (Vd) of [14C]GSK1120212 and total drug-related material (radioactivity)
AEs | Day 1, Day 2, Day 3, Day 4, Day 6, Day 8, Day 11, and follow-up.
  Number of AEs
Blood pressure | Screening, Day 1, Day 2, and follow-up.
  Change from baseline
Pulse rate | Screening, Day 1, Day 2, and follow-up.
  Change from baseline
ECG | Screening, Day 1, Day 2, and follow-up.
  Change from baseline
Echo | Screening day and follow-up
  Change from baseline
Clinical Laboratory data | Screening, Day 1, and follow-up.
  Change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tacoma, Washington, United States

REFERENCES:
- [Derived] Leonowens C, Pendry C, Bauman J, Young GC, Ho M, Henriquez F, Fang L, Morrison RA, Orford K, Ouellet D. Concomitant oral and intravenous pharmacokinetics of trametinib, a MEK inhibitor, in subjects with solid tumours. Br J Clin Pharmacol. 2014 Sep;78(3):524-32. doi: 10.1111/bcp.12373. PMID 24606567
- See also: Results for study 115064 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115064?search=study&study_ids=115064#rs